CLINICAL TRIAL: NCT04202757
Title: Intravenous Young Fresh Frozen Plasma (yFFP) Investigational Treatment for Parkinson's Disease
Brief Title: Intravenous Plasma Treatment for Parkinson's Disease
Acronym: yFFP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Neurology Center (Other)
Collaborators: Carolina Longevity Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NeurologyCenter
Record Dates: First submitted 2018-09-21; First posted 2019-12-18 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Placebo controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinding will be achieved by preparing both yFFP and placebo (0.1% riboflavin in normal saline) solution into identical-sized, masked bags. The riboflavin is added to the saline to achieve indistinguishable color when compared to the yFFP. Physicians who evaluate patients are masked from treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Young Fresh Frozen Plasma (yFFP) (Active Comparator): [21CFR640.30] Plasma from 18 - 25 year old volunteer donors
  Interventions: Biological: [21CFR640.30] Plasma from 18 - 25 year old volunteer donors
- Saline (Placebo Comparator): 0.1% riboflavin in normal saline
  Interventions: Other: Saline

INTERVENTIONS:
Biological: [21CFR640.30] Plasma from 18 - 25 year old volunteer donors — 12.5 ml/kg intravenous Spectrum Plasma yFFP, per each of two infusions (25 ml/kg total), in combination with ongoing normal standard treatment.
  Other Names: Young Fresh Frozen Plasma (yFFP)
  Arms: Young Fresh Frozen Plasma (yFFP)
Other: Saline — 12.5 ml/kg intravenous 0.9% sodium chloride with 0.1% riboflavin , per each of two infusions (25 ml/kg total), in combination with ongoing normal standard treatment.
  Other Names: Normal saline
  Arms: Saline

SUMMARY:
This study will do a preliminary evaluation of a possible treatment for mild-to-moderate Parkinson's disease. Patients will be treated with either transfusions of plasma from young donors. or with placebo transfusions. In the following several months, Parkinson's symptoms will be monitored and compared for the two groups.

DETAILED DESCRIPTION:
This is a double-blind placebo controlled trial, designed to evaluate the efficacy of plasma from volunteer donors of ages 18-25. This young fresh frozen plasma (yFFP) will be given intravenously in two doses of 12.5 ml/kg each, with 40-56 hours between doses. In the following 24 weeks, Parkinson's symptoms will be monitored using the short version of the Stanford Presenteeism Scale (SPS-6), and a modified version of the UPDRS scale.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* Disease duration of 1 to 5 years
* Willingness to confirm the use of adequate birth control while on the trial will be required in premenopausal women without evidence for an inability to become pregnant.
* Willingness to not start any other treatment for Parkinson's or Multiple Sclerosis during the parallel part of the trial.

Exclusion Criteria:

* Other significant disease, which in the view of the study doctor may make assessment of the efficacy of yFFP difficult.
* Unstable medical conditions.
* Must weigh at least 45.5 kg. Cannot weigh more than 130 kg.
* A severe disease state diagnosis
* Litigation. Patients in litigation will be excluded only if conclusion of that litigation is imminent during the course of the study.
* If patient is pregnant or breastfeeding.
* Complete IgA deficiency.
* Rare contraindications to yFFP therapy as per summary of product characteristics.
* Receiving yFFP for other reasons.
* Ongoing drug or alcohol abuse.
* Psychiatric disorder that could, in the judgement of the site investigator, interfere with successful study participation.
* Unwillingness or inability to complete the study or an inability to understand the questionnaires being used.
* Cancer other than basal cell carcinoma within the last 5 years. However, those patients who have received definitive treatment, such as curative surgery more than 6 months ago, with no known recurrence can be included.
* A history of hypercoagulable or thrombophilic clotting abnormalities.
* A history of thromboembolic events: ischaemic stroke, confirmed myocardial infarction, pulmonary embolism; deep venous thrombosis except where immobility related (for example, after injury or operation).
* Unstable angina pectoris.
* Medications that might react with yFFP such as blood thinners
* Renal failure or serum creatinine greater than 1.5 times the upper limit of normal at screening.
* Any medical condition that, in the opinion of the investigator, would make it unsafe for the patient to participate or which would interfere with assessment of the outcome measures.
* Participation in another interventional trial within 3 months of randomization. Participation in non-interventional studies is not a reason for exclusion.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Changes in Physician assessment | Two weeks prior to infusion, at one-three-six months post-infusion
  Unified Parkinson Disease Rating Scale (UPDRS)
Patient assessment | Two weeks prior to infusion, at one-three-six months post-infusion
  Changes in Stanford Presenteeism Scale (SPS)

SECONDARY OUTCOMES:
Stability of administration | At the time of infusions, day 1 and day 2
  Adverse events (if any)
Factors predicting a beneficial response | After the last participant's final contact at 6 months
  Patient Global Impression of change

CONTACTS AND LOCATIONS:
Overall Officials: Dian Ginsberg, M.D., Principal Investigator — The Ginstitute of Functional Medicine
Locations (1):
- The Neurology Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT04202757/Prot_SAP_002.pdf
  • Informed Consent Form (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT04202757/ICF_003.pdf